CLINICAL TRIAL: NCT06541717
Title: Midwifery Students' Ovarian Reserve and Fertility Awareness: Effectiveness of Video Intervention
Brief Title: Video Intervention Fertility Awareness Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-008
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Video-Based Fertility Awareness Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:40) (Experimental): Students will be shown 3 15-minute videos created by researchers on the anatomy and physiology of the male and female reproductive systems, the physiology of pregnancy, fertility awareness development and its importance in terms of infertility.
  Interventions: Other: Video-Based Fertility Awareness Training
- Control group (n:40) (No Intervention): Students will be trained for 2 hours using the classical method on the anatomy and physiology of the male and female reproductive systems, the physiology of pregnancy, fertility awareness development and its importance in terms of infertility.

INTERVENTIONS:
Other: Video-Based Fertility Awareness Training — Students will be shown 3 15-minute videos created by researchers on the anatomy and physiology of the male and female reproductive systems, the physiology of pregnancy, fertility awareness development and its importance in terms of infertility.
  Arms: İntervention group (n:40)

SUMMARY:
This study was planned to evaluate the effects of video-based ovarian reserve awareness training applied to midwifery students on ovarian reserve, fertility awareness and anxiety of midwifery students. The research population will consist of second-year students studying in the Department of Midwifery, Hamidiye Faculty of Health Sciences (HSBF), Health Sciences University (SBU) in the fall semester of 2024-2025 academic year (N: 80). In this study planned as a semi-experimental pre-test and post-test design with a control group, in order to determine the sample size; the data were normally distributed, the standard deviation of the main mass was estimated as 1 and the effect size (effect size, difference) was estimated as 0.8. For the analysis to be conducted, it was calculated that the highest power value of the study would be 0.942182 if two independent n₁=40, n₂=40 samples were taken at a significance level of 5%. The G-power analysis result is given below.

Students who volunteer to participate in the study will be assigned to the intervention and control groups with the computer-aided simple random sampling method. Computer-aided randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www.randomizer.org and random assignment will be made to the intervention and control groups. The study will be conducted single-blind. Midwifery students in the intervention group of the study will be given video-based ovarian reserve and fertility awareness training. A pre-training information meeting will be held with midwifery students who volunteered to participate in the study and were assigned to the intervention group. The midwifery students will be administered the "Ovarian Reserve Information Form", "Fertility Awareness Scale" and "State Anxiety Scale" before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* To be a volunteer to participate in the research.
* To be an active student in the 2nd year of the Midwifery Department of Hamidiye Health Sciences Faculty, University of Health Sciences.

Exclusion Criteria:

* Being a passive student in the 2nd year of the Midwifery Department of Hamidiye Health Sciences Faculty, University of Health Sciences.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  It was prepared by the researchers after conducting a literature research and taking expert opinions. The form includes questions about the sociodemographic characteristics of the students.
Ovarian Reserve Information Form | 10 minutes
  It was prepared by researchers after conducting a literature review and obtaining expert opinions. The form includes questions that evaluate students' knowledge and attitudes about ovarian reserve.
Fertility Awareness Scale (FAS) | 10 minutes
  The Fertility Awareness Scale (FAS) is a Likert-type scale consisting of 19 items and two dimensions. There is no reverse item in the scale. The lowest score that can be obtained from the FAS is 19 and the highest score is 95. The range is 10-50 in the Physical Awareness sub-dimension and 9-45 in the Cognitive Awareness sub-dimension. As the total score obtained from the FAS increases, the level of awareness increases. When evaluating the total score obtained from the FAS; if the total score is between 19-43, awareness is scored as low, if it is between 44-69, awareness is scored as medium, and if it is between 70-95, awareness is scored as high. These values were determined according to the calculation of the score range average method. Cronbach's alpha internal consistency coefficient was determined as 0.887 for the total FAS scale.
State-Trait Anxiety Inventory | 10 minutes
  This inventory, developed by Spielberger et al. (1970), consists of two subscales, state and trait, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how an individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how an individual feels independently of the situation and conditions they are in. The adaptation of the State and Trait Anxiety Inventory to Turkish, its validity and reliability study was conducted by Öner and Le Compte (1983).

SECONDARY OUTCOMES:
Ovarian Reserve Information Form | 10 minutes
  It was prepared by researchers after conducting a literature review and obtaining expert opinions. The form includes questions that evaluate students' knowledge and attitudes about ovarian reserve.
Fertility Awareness Scale (FAS) | 10 minutes
  The Fertility Awareness Scale (FAS) is a Likert-type scale consisting of 19 items and two dimensions. There is no reverse item in the scale. The lowest score that can be obtained from the FAS is 19 and the highest score is 95. The range is 10-50 in the Physical Awareness sub-dimension and 9-45 in the Cognitive Awareness sub-dimension. As the total score obtained from the FAS increases, the level of awareness increases. When evaluating the total score obtained from the FAS; if the total score is between 19-43, awareness is scored as low, if it is between 44-69, awareness is scored as medium, and if it is between 70-95, awareness is scored as high. These values were determined according to the calculation of the score range average method. Cronbach's alpha internal consistency coefficient was determined as 0.887 for the total FAS scale.
State-Trait Anxiety Inventory | 10 minutes
  This inventory, developed by Spielberger et al. (1970), consists of two subscales, state and trait, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how an individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how an individual feels independently of the situation and conditions they are in. The adaptation of the State and Trait Anxiety Inventory to Turkish, its validity and reliability study was conducted by Öner and Le Compte (1983).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No